CLINICAL TRIAL: NCT03381300
Title: Preservation of Ovarian Cortex Tissue in Girls With Turner Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL57738.000.16
Record Dates: First submitted 2017-11-22; First posted 2017-12-21 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Fertility Preservation; Ovarian Tissue Cryopreservation; Turner Syndrome; Live Birth; Premature Ovarian Failure
MeSH Terms: conditions — Turner Syndrome; Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single cohort (Other)
  Interventions: Procedure: Ovarian tissue cryopreservation

INTERVENTIONS:
Procedure: Ovarian tissue cryopreservation — Laparoscopic unilateral oophorectomy followed by cryopreservation of ovarian cortex tissue

SUMMARY:
Rationale: Infertility due is a major concern for girls with Turner syndrome (TS) and their parents. Physicians are often asked about possible options to preserve their fertility. However, despite some experimental case reports, clear evidence for fertility preservation in these girls is lacking and many questions remain. Without evidence on the effectiveness of fertility preservation it cannot routinely be offered to girls with TS.

Objective: To investigate the occurrence of live birth in women with TS after ovarian tissue cryopreservation in childhood followed by auto transplantation in adulthood.

Study design: A national multicentre exploratory intervention study

Study population: Girls diagnosed with Turner Syndrome, aged 2-18 years.

Intervention: Ovarian tissue cryopreservation in childhood followed by auto transplantation in adulthood. In order to obtain the ovarian tissue for cryopreservation, all girls must undergo a laparoscopy under general anaesthesia which will be performed in academic/university clinics with paediatric surgery. During the laparoscopic intervention, a unilateral oophorectomy will be performed, thereby leaving the other ovary intact for hormone production, ovulation, spontaneous pregnancies and as an auto transplantation site for cryopreserved-thawed ovarian cortical tissue later on. Furthermore, a small sample of the ovarian cortex will be used to assess the oocyte quality and genetics (e.g. the presence of germ line mosaicism). Oocytes will be karyotyped by using Fluorescence in situ hybridization (FISH). Karyotypic and hormonal data will be collected once at the yearly clinical visit at the paediatric-endocrinologist. Therefore, a buccal swab and one extra blood sample will be taken and evaluated during the routine laboratory evaluation.

In the future, auto transplantation of frozen-thawed ovarian cortex strips will be performed.

DETAILED DESCRIPTION:
Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The primary objective remains to preserve the fertility of the respective (minor) patient, facing a very high risk of premature ovarian insufficiency (POI) of 95-98%. Disadvantages of participating in this study are the potential risk of complications related to the laparoscopic unilateral oophorectomy and/or the unknown effect on future fertility of these girls. Moreover, the procedure might raise false hope in patients (and/or parents) about the chance of getting pregnant after auto transplantation of cryopreserved-thawed ovarian tissue in the future. However, we attempt to overcome this by extensive and objective information provision by both written materials and face to face counselling.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Girls and young females with classic Turner (i.e. 45X monosomy) or Turner variants (e.g. 45X / 46XX mosaicism, ring X mosaicism, isochromosome X),
* Aged 2 through 18 years,
* who completed the diagnostic work up phase of TS including routine cardiac screening*,
* whose agreement to participate in this study has been signed by the parents (girls 2-11 years old),
* whose agreement to participate in this study has been signed by the patient and her parents (girls 12-17 years old),
* whose agreement to participate in this study has been signed by the patient (adolescents of 18 years old).

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Contra-indications for laparoscopic unilateral oophorectomy under general anaesthesia (e.g. severe cardiovascular comorbidity and/or BMI >40 kg/m2)*,
* Contra-indications for cryopreservation (i.e. active HIV, hepatitis-B or hepatitis-C infection)

  * Based on the international Cincinnati Turner Guideline consensus Meeting, July 2016 and consultation of Dutch cardiologists, paediatric-cardiologists and anaesthesists between 2016-2017 there are no absolute cardiovascular contra-indications for surgical intervention and/or pregnancy. Advice against surgical intervention and/or pregnancy should be based on the patient-specific cardiovascular risk profile. The 2% mortality risk due to acute aortic dissection is based on one survey and literature review study that reported the outcomes of 101 pregnancies in patients with TS after oocyte donation. Only 50% of the patients were screened by a cardiologist before entering the oocyte donation programme. Therefore, all girls who want to participate in this study should have completed the diagnostic work up phase of TS including routine cardiac screening and will be screened by a paediatric anaesthesist. Exclusion will be based on the patient specific risk profile. See: References.

Ages: 2 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Patients 45X monosomy of mosaicism
Enrollment: 106 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2071-11-01 (Estimated); Study Completion 2071-11-01 (Estimated)

PRIMARY OUTCOMES:
Live birth ratio (LBR) (main outcome) | Up to 3 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue, and up to 45 years after ovarian tissue cryopreservation.
  • Live birth after auto transplantation of cryopreserved-thawed ovarian cortical tissue (i.e. live birth rate or LBR)
Number of primordial follicles (proximate) | Within 1 month after ovarian tissue cryopreservation
  The number of primordial follicles found in the ovarian tissue

SECONDARY OUTCOMES:
Patient's age versus LBR | Up to 3 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue, and up to 45 years after ovarian tissue cryopreservation.
  The association between patient's age at cryopreservation and LBR
Patient's genotype versus LBR | Up to 3 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue, and up to 45 years after ovarian tissue cryopreservation.
  The association between patient's genotype and LBR
Patient's Anti-Müllerian hormone (AMH) level versus LBR | Up to 3 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue, and up to 45 years after ovarian tissue cryopreservation.
  The association between patient's AMH level at cryopreservation and LBR
Patient's Follicle-stimulating hormone (FSH) level versus LBR | Up to 3 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue, and up to 45 years after ovarian tissue cryopreservation.
  The association between patient's FSH level at cryopreservation and LBR

OTHER OUTCOMES:
Study participation rate | Up to 3 years after inclusion
  The willingness of girls with TS to perform a unilateral oophorectomy for fertility preservation (i.e. the study participation rate)
Eligible participants | Up to 3 years after inclusion
  The number of eligible participants
Age | Up to 3 years after inclusion
  The age of the participant
Buccal cells versus peripheral lymphocytes | Up to 3 years after inclusion
  The incidence of somatic mosaicism (i.e. buccal cells versus peripheral lymphocytes)
Ovarian cells versus peripheral lymphocytes | Up to 3 years after inclusion
  The incidence of germ cell mosaicism (i.e. ovarian cells versus peripheral lymphocytes and buccal cells)
Serum hormone levels | Up to 3 years after inclusion
  Serum hormone levels (i.e. FSH, Luteinizing hormone (LH), AMH, E2, inhibin B)
Complication rate | Up to 1 year after the laparoscopic procedure
  The number of complications related to the laparoscopic procedure
Influence of laparoscopic oophorectomy on puberty and/or menarche | Up to 10 years after the laparoscopic procedure
  The incidence of puberty and/or menarche after laparoscopic oophorectomy
Incidence of spontaneous pregnancies | Up to 45 years after the laparoscopic procedure
  The incidence of spontaneous pregnancies after laparoscopic oophorectomy
Restoration of ovarian function after auto transplantation of ovarian tissue | Up to 2 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue
  The incidence of menstruation cycle recovery after auto transplantation of cryopreserved-thawed ovarian tissue in the future
Pregnancies after auto transplantation of ovarian tissue | Up to 2 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue
  The incidence of pregnancies after auto transplantation of cryopreserved-thawed ovarian tissue in the future
Ongoing pregnancies after auto transplantation of ovarian tissue | Up to 2 years and 3 months after auto transplantation of cryopreserved-thawed ovarian cortical tissue
  The incidence of ongoing pregnancies after auto transplantation of cryopreserved-thawed ovarian tissue in the future
Miscarriages after auto transplantation of ovarian tissue | Up to 3 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue
  The number of miscarriages after auto transplantation of cryopreserved-thawed ovarian tissue in the future
Time to pregnancy after auto transplantation of ovarian tissue | Up to 2 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue
  Time to pregnancy after auto transplantation of cryopreserved-thawed ovarian tissue in the future
Time to live birth after auto transplantation of ovarian tissue | Up to 3 years after auto transplantation of cryopreserved-thawed ovarian cortical tissue
  Time to live birth after auto transplantation of cryopreserved-thawed ovarian tissue in the future

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Fleischer, MD, PhD, Principal Investigator — Head Department of Reproductive Medicine, Gynaecologist/Subspecialist Reproductive Medicine
Locations (1):
- Radboud university medical center. Department Obstetrics & Gynaecology., Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gravholt CH, Andersen NH, Conway GS, Dekkers OM, Geffner ME, Klein KO, Lin AE, Mauras N, Quigley CA, Rubin K, Sandberg DE, Sas TCJ, Silberbach M, Soderstrom-Anttila V, Stochholm K, van Alfen-van derVelden JA, Woelfle J, Backeljauw PF; International Turner Syndrome Consensus Group. Clinical practice guidelines for the care of girls and women with Turner syndrome: proceedings from the 2016 Cincinnati International Turner Syndrome Meeting. Eur J Endocrinol. 2017 Sep;177(3):G1-G70. doi: 10.1530/EJE-17-0430. PMID 28705803
- [Derived] van der Coelen S, Nadesapillai S, Peek R, Braat D, Bocca G, Finken M, Hannema S, de Kort S, Sas T, Straetemans S, van Tellingen V, Stuart AV, Fleischer K, van der Velden J. Puberty progression in girls with Turner syndrome after ovarian tissue cryopreservation. Fertil Steril. 2025 Apr;123(4):583-592. doi: 10.1016/j.fertnstert.2024.10.025. Epub 2024 Oct 19. PMID 39433199
- [Derived] Nadesapillai S, van der Velden J, van der Coelen S, Schleedoorn M, Sedney A, Spath M, Schurink M, Oerlemans A, IntHout J, Beerendonk I, Braat D, Peek R, Fleischer K. TurnerFertility trial: fertility preservation in young girls with Turner syndrome by freezing ovarian cortex tissue-a prospective intervention study. Fertil Steril. 2023 Nov;120(5):1048-1060. doi: 10.1016/j.fertnstert.2023.08.004. Epub 2023 Aug 5. PMID 37549836
- [Derived] Nadesapillai S, van der Velden J, Smeets D, van de Zande G, Braat D, Fleischer K, Peek R. Why are some patients with 45,X Turner syndrome fertile? A young girl with classical 45,X Turner syndrome and a cryptic mosaicism in the ovary. Fertil Steril. 2021 May;115(5):1280-1287. doi: 10.1016/j.fertnstert.2020.11.006. Epub 2020 Dec 17. PMID 33342535
- [Derived] Schleedoorn M, van der Velden J, Braat D, Beerendonk I, van Golde R, Peek R, Fleischer K. TurnerFertility trial: PROTOCOL for an observational cohort study to describe the efficacy of ovarian tissue cryopreservation for fertility preservation in females with Turner syndrome. BMJ Open. 2019 Dec 11;9(12):e030855. doi: 10.1136/bmjopen-2019-030855. PMID 31831533
- [Derived] Peek R, Schleedoorn M, Smeets D, van de Zande G, Groenman F, Braat D, van der Velden J, Fleischer K. Ovarian follicles of young patients with Turner's syndrome contain normal oocytes but monosomic 45,X granulosa cells. Hum Reprod. 2019 Sep 29;34(9):1686-1696. doi: 10.1093/humrep/dez135. PMID 31398245

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT03381300/Prot_SAP_000.pdf